CLINICAL TRIAL: NCT05119062
Title: The Feasibility of an Online Intergenerational Co-parenting Program for Father-mother-grandmother Triad on the Intergenerational Co-parenting Relationship in the Perinatal Period
Brief Title: The Feasibility of an Online Intergenerational Co-parenting Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Shenzhen Maternity & Child Healthcare Hospital (Other)
Responsible Party: Principal Investigator, Ngai Fei Wan, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSEARS20210927005
Record Dates: First submitted 2021-10-22; First posted 2021-11-12 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Intergenerational Relations; Perinatal Depression; Parenting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): Participants in the control group will receive usual care.
  Interventions: Other: Usual care
- an online intergenerational co-parenting programme (Experimental): Those who are randomized to the intervention group will receive the intergenerational co-parenting program in addition to the usual care, including 3 weekly antenatal sessions (start from 33-35 weeks gestation) and 2 weekly postnatal sessions (start from the first week after discharge from hospital). The essential components and focus of the intergenerational co-parenting program were developed based on the themes identified from the two qualitative studies, the systematic review of co-parenting interventions, and the proposed intergenerational co-parenting model. The intervention will be delivered online through an education platform of the study hospital.
  Interventions: Other: an online intergenerational co-parenting programme+usual care

INTERVENTIONS:
Other: Usual care — Families in the control group will be provided with routine care, including regular antenatal check ups, one bed side education (within 24 hours after delivery), one group session with discharge precautions (3rd to 5th day postpartum), two home visits (first week and second week after discharge respectively), and two physical body check at hospital on the 30th and 42nd day postpartum. Contents of the bed side education, pre-discharge education and home visits focuses on health related information, such as postpartum care, infant care and breastfeeding, etc.
  Arms: Control group
Other: an online intergenerational co-parenting programme+usual care — The program is proposed to include five sessions, with three antenatal sessions to be offered weekly during the 34-36 weeks gestation and two postnatal sessions weekly starting from the first week after discharge from hospital. The intervention will be delivered online.The program is designed for the intergenerational co-parenting families to undertake with parents together with grandmothers. The online courses will be delivered by an online platform in the study hospital. The first session will be pushed to participants in the intervention group within 2 days (around 34 weeks gestation) after recruitment. The second and third session will be pushed around 35 and 36 weeks gestation separately. The first postnatal session will be provided around the first to second week postpartum; and second postnatal session will be provided around the third to fourth week postpartum.
  Arms: an online intergenerational co-parenting programme

SUMMARY:
This is a feasibility study with pilot randomized controlled trial design. A convenience sample of 60 intergenerational co-parenting family units, including 60 first-time parents (60 mothers and 60 fathers) and 60 grandmothers (mother-in-law of mothers) will be recruited from the obstetric clinics in the outpatient department of the study hospital, with 30 family units of each in the intervention group and control group respectively. Participants who are recruited will be randomly assigned to the intervention or control group by a research assistant based on the sequential enrollment list. Participants in the control group will receive usual care. Those who are randomized to the intervention group will receive the intergenerational co-parenting program in addition to the usual care.

DETAILED DESCRIPTION:
This is a feasibility study with pilot randomized controlled trial design. A convenience sample of 60 intergenerational co-parenting family units, including 60 first-time parents (60 mothers and 60 fathers) and 60 grandmothers (mother-in-law of mothers) will be recruited from the obstetric clinics in the outpatient department of the study hospital, with 30 family units of each in the intervention group and control group respectively. A sequential enrollment list linked to a random number sequence will be generated by a statistician. Participants who are recruited will be randomly assigned to the intervention or control group by a research assistant based on the sequential enrollment list. Participants in the control group will receive usual care. Those who are randomized to the intervention group will receive the intergenerational co-parenting program in addition to the usual care, including 3 weekly antenatal sessions (start from 33-35 weeks gestation) and 2 weekly postnatal sessions (start from the first week after discharge from hospital). The essential components and focus of the intergenerational co-parenting program were developed based on the themes identified from the two qualitative studies, the systematic review of co-parenting interventions, and the proposed intergenerational co-parenting model. The intervention will be delivered online through an education platform of the study hospital. The acceptability, feasibility of the intergeneration co-parenting program will be examined. In addtion, the preliminary effects of such program on the intergenerational co-parenting relationship between mothers and grandmothers reported by mothers (primary outcome), and on the secondary outcomes: the psychological well-being of parents and grandmothers, the co-parenting relationship between parents, parenting stress and parenting self-efficacy of parents at 6 weeks, and 3 months postpartum will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* the inclusion criteria for this study will be: (1) first time expectant parents (at least 18 years old) and should be married couples; (2) women have no pregnancy complications and around 34 weeks gestation (33-35 weeks); (3) women have regular antenatal check-ups in the study hospital and are going to deliver in the study hospital; (4) women living in Shenzhen together with husband, is cared by their mother-in-law at recruitment and will be taken care of by their mother-in-law in Shenzhen during the postpartum period; (5) Both parents and grandmothers could understand, read and speak mandarin and are willing to take part in this study; (6) Both parents and grandmothers are able to use smart phone and know how to use Wechat since the message from the online platform is pushed to Wechat in this study.

Exclusion Criteria:

* Intergeneration coparenting families will be excluded if members of the family unit with reported mental health problems, such as schizophrenia, bipolar affective disorders, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
intergenerational co-parenting relationship | 6 weeks postpartum
  The Chinese version of Co-parenting relationship Scale (Feinberg et al., 2012; Li & Wei, 2018) will be used to assess the intergenerational co-parenting relationship between mothers and grandmothers reported by mothers. There are 38 items in the Chinese version of CRS. The total score ranges from 38 to 266. The Exploratory Factor Analysis adopted 7 factors. The internal consistency ranged from 0.65 to 0.87, the split half reliability was 0.60 to 0.86, and the test-retest reliability was 0.38 to 0.71. Higher scores indicate better intergenerational co-parenting relationship.
intergenerational co-parenting relationship | 3 months postpartum
  The Chinese version of Co-parenting relationship Scale (Feinberg et al., 2012; Li & Wei, 2018) will be used to assess the intergenerational co-parenting relationship between mothers and grandmothers reported by mothers. There are 38 items in the Chinese version of CRS. The total score ranges from 38 to 266. The Exploratory Factor Analysis adopted 7 factors. The internal consistency ranged from 0.65 to 0.87, the split half reliability was 0.60 to 0.86, and the test-retest reliability was 0.38 to 0.71. Higher scores indicate better intergenerational co-parenting relationship.

SECONDARY OUTCOMES:
The depressive symptoms of co-parenting members | baseline at around 33-35 weeks gestation
  The Center for Epidemiological Studies Depression Scale (Radloff, 1977) will be used. The scale contains 20 items. The participants are asked to recall the symptoms that they experienced during the past week and respond with answers on a 4-point frequency. Each item is scored from 0 to 3, with total scores ranging from 0 to 60. A higher score indicates greater depression.
The depressive symptoms of co-parenting members | 6 weeks postpartum
  The Center for Epidemiological Studies Depression Scale (Radloff, 1977) will be used. The scale contains 20 items. The participants are asked to recall the symptoms that they experienced during the past week and respond with answers on a 4-point frequency. Each item is scored from 0 to 3, with total scores ranging from 0 to 60. A higher score indicates greater depression.
The depressive symptoms of co-parenting members | 3 months postpartum
  The Center for Epidemiological Studies Depression Scale (Radloff, 1977) will be used. The scale contains 20 items. The participants are asked to recall the symptoms that they experienced during the past week and respond with answers on a 4-point frequency. Each item is scored from 0 to 3, with total scores ranging from 0 to 60. A higher score indicates greater depression.
The perceived stress of co-parenting members | baseline at around 33-35 weeks gestation
  The short version of Perceived Stress Scale-4 (Cohen, 1983) will be to assess the perceived stress of co-parenting members. It consists of 4 items. Respondents rate each item with the frequency with which they experienced stress in the last month, ranging from 0 (never) to 4 (very often). The total score rangs from 0 to 16. Higher scores indicate that the respondents suffer from greater stress.
The perceived stress of co-parenting members | 6 weeks postpartum
  The short version of Perceived Stress Scale-4 (Cohen, 1983) will be to assess the perceived stress of co-parenting members. It consists of 4 items. Respondents rate each item with the frequency with which they experienced stress in the last month, ranging from 0 (never) to 4 (very often). The total score rangs from 0 to 16. Higher scores indicate that the respondents suffer from greater stress.
The perceived stress of co-parenting members | 3 months postpartum
  The short version of Perceived Stress Scale-4 (Cohen, 1983) will be to assess the perceived stress of co-parenting members. It consists of 4 items. Respondents rate each item with the frequency with which they experienced stress in the last month, ranging from 0 (never) to 4 (very often). The total score rangs from 0 to 16. Higher scores indicate that the respondents suffer from greater stress.
Co-parenting relationship between couples | 6 weeks postpartum
  The Chinese version of The brief Co-parenting Relationship Scale (Feinberg et al., 2012; Wu, Li & Zhao, 2017) will be used to assess the co-parenting relationship between couples. The scale contains 14 items covering seven domains. Each item is rated on a 7-point Likert Scale from 0 to 6, with total scores ranging from 0 to 84. The Cronbach's alpha of Chinese version is 0.613, and the exploratory factor analysis showed Model fit was acceptable, with a reported KMO 0.748, Bartlett's χ2=686.086, P<0.01.
Co-parenting relationship between couples | 3 months postpartum
  The Chinese version of The brief Co-parenting Relationship Scale (Feinberg et al., 2012; Wu, Li & Zhao, 2017) will be used to assess the co-parenting relationship between couples. The scale contains 14 items covering seven domains. Each item is rated on a 7-point Likert Scale from 0 to 6, with total scores ranging from 0 to 84. The Cronbach's alpha of Chinese version is 0.613, and the exploratory factor analysis showed Model fit was acceptable, with a reported KMO 0.748, Bartlett's χ2=686.086, P<0.01.
Parenting stress of parents | 6 weeks postpartum
  The parenting stress of parents will be measured using the Short Version of the Parenting Stress Index (Abidin & Abidin, 1990). The subscale of parental distress (PD) (12 items) and parent-child dysfunctional interaction (PCDI) (12 items) will be used in this study (Leung et al., 2005; Liu, Chen, Yeh, & Hsieh, 2012). The content validity of the Chinese version was 0.86 and the reliability was 0.91 after the removal of the DC subscale (Liu et al., 2012). Respondents are asked to rate the items using a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Total scores of these two subscales range from 24 to 120, with scores ranging from 12 to 60 for each subscale (Liu et al., 2012). A higher score predicts higher parenting stress.
Parenting stress of parents | 3 months postpartum
  The parenting stress of parents will be measured using the Short Version of the Parenting Stress Index (Abidin & Abidin, 1990). The subscale of parental distress (PD) (12 items) and parent-child dysfunctional interaction (PCDI) (12 items) will be used in this study (Chan et al., 2005; Liu, Chen, Yeh, & Hsieh, 2012). The content validity of the Chinese version was 0.86 and the reliability was 0.91 after the removal of the DC subscale (Liu et al., 2012). Respondents are asked to rate the items using a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Total scores of these two subscales range from 24 to 120, with scores ranging from 12 to 60 for each subscale (Liu et al., 2012). A higher score predicts higher parenting stress.
Parenting self-efficacy of parents | 6 weeks postpartum
  The Parenting Sense of Competence Scale (Gibaud-Wallston & Wandersman, 2001) will be used to assess the parenting self-efficacy of parents. This 17-item scale consists of two subscales, and has been widely used for assessments of parenting self-efficacy. Each item is rated from 1 to 6, with a total socre ranging from 17 to 102. A higher score indicates higher parenting self-efficacy. The Cronbach's alpha was 0.85 for the total scale in the Chinese version, and 0.80 and 0.77 for the subscales of Efficacy and Satisfaction, respectively. The test-retest reliability was 0.87. Good construct validity was also confirmed in the Chinese version via factor analyses, where 82% of the factors were loaded (Ngai, Chan, & Holroyd, 2007).
Parenting self-efficacy of parents | 3 months postpartum
  The Parenting Sense of Competence Scale (Gibaud-Wallston & Wandersman, 2001) will be used to assess the parenting self-efficacy of parents. This 17-item scale consists of two subscales, and has been widely used for assessments of parenting self-efficacy. Each item is rated from 1 to 6, with a total socre ranging from 17 to 102. A higher score indicates higher parenting self-efficacy. The Cronbach's alpha was 0.85 for the total scale in the Chinese version, and 0.80 and 0.77 for the subscales of Efficacy and Satisfaction, respectively. The test-retest reliability was 0.87. Good construct validity was also confirmed in the Chinese version via factor analyses, where 82% of the factors were loaded (Ngai, Chan, & Holroyd, 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Ngai Feiwan, PhD, Principal Investigator — School of Nursing
Locations (2):
- China (2):
  - Shenzhen Maternity & Child Healthcare Hospital, Shenzhen, Guangdong
  - Hong Kong Polytechnic University, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abidin, R. R., & Abidin, R. R. (1990). Parenting Stress Index (PSI)(p. 100).
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Feinberg ME, Brown LD, Kan ML. A Multi-Domain Self-Report Measure of Coparenting. Parent Sci Pract. 2012 Jan 1;12(1):1-21. doi: 10.1080/15295192.2012.638870. Epub 2012 Jan 20. PMID 23166477
- [Background] Gibaud-Wallston, J., & Wandersman, L. (2001). Parenting sense of competence scale (PSOC).
- [Background] Li, X.W., & Wei, X.Y. (2018). Revision of the Grandparents-Parents Co-parenting Relationships Scale in Chinese Families. Chinese Journal of Clinical Psychology, 26(5):882-886. In Chinese.
- [Background] Radloff, L. S. (1977). The CES-D scale: A self-report depression scale for research in the general population. Applied Psychological Measurement, 1(3), 385-401.
- [Background] Wu, J.M., Li, G.J. & Zhao, H. (2017). Reliability and validity of the Chinese version of the Brief co-parenting Relationship Scale. Research on Maternal and Child Health in China, 28 (4), 369-371. In Chinese
- [Background] Liu CC, Chen YC, Yeh YP, Hsieh YS. Effects of maternal confidence and competence on maternal parenting stress in newborn care. J Adv Nurs. 2012 Apr;68(4):908-18. doi: 10.1111/j.1365-2648.2011.05796.x. Epub 2011 Jul 27. PMID 21790741
- [Background] Ngai FW, Wai-Chi Chan S, Holroyd E. Translation and validation of a chinese version of the parenting sense of competence scale in chinese mothers. Nurs Res. 2007 Sep-Oct;56(5):348-54. doi: 10.1097/01.NNR.0000289499.99542.94. PMID 17846556
- [Background] Leung C, Leung S, Chan R, Tso K, Ip F. Child behaviour and parenting stress in Hong Kong families. Hong Kong Med J. 2005 Oct;11(5):373-80. PMID 16219957